CLINICAL TRIAL: NCT01516931
Title: A Study to Evaluate the Efficacy of Repetitive Transcranial Magnetic Stimulation in the Prevention of Relapse of the Symptoms of Depression.
Brief Title: Efficacy of Repetitive Transcranial Magnetic Stimulation in the Prevention of Relapse of Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Collaborators: The No.3 hospital of PLA (Unknown); The No.91 hospital of PLA (Unknown); No. 102 Hospital of Chinese People's Liberation Army (Other)
Responsible Party: Principal Investigator, Huaning Wang, director of department, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Huaning Wang; XijingH (Other: XijingH)
Record Dates: First submitted 2011-12-29; First posted 2012-01-25 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Depression
Keywords: repetitive Transcranial Magnetic Stimulation (rTMS); Depression; Venlafaxine; Relapse
MeSH Terms: conditions — Depression; Recurrence | interventions — Transcranial Magnetic Stimulation; Counseling

STUDY DESIGN:
Intervention Model Description: rTMS intervention
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- active rTMS and venlafaxine (Experimental): rTMS：Intensity of 120% of individually determined motor threshold; frequency : 1 Hz; 360 impulsions; on period : 1 min; off period : 30 s.5 sessions per week for 4-6 weeks,than 2 sessions per week for 2 months, repeat that for 12 months.
  venlafaxine：150-225mg/day
  Interventions: Procedure: repetitive Transcranial Magnetic Stimulation (rTMS)
- sham rTMS and venlafaxine (Placebo Comparator): Sham stimulation will be given at the same site and frequency, using a Magstim sham-coil system. During rTMS, participants will be instructed to keep their eyes open and relax.
  Interventions: Behavioral: counseling
- venlafaxine alone (Placebo Comparator): responders will be maintained on the same effective dose of venlafaxine for the entire duration of the RCT, unless they relapse and will have to exit the protocol and enter a naturalistic follow-up
  Interventions: Behavioral: counseling

INTERVENTIONS:
Procedure: repetitive Transcranial Magnetic Stimulation (rTMS) — 1 Hz; 360 impulsions; on period : 1 min; off period : 30 s.5 sessions per week for 4-6 weeks
  Arms: active rTMS and venlafaxine
Behavioral: counseling — Placebo monthly by general counseling for 12 months.
  Arms: sham rTMS and venlafaxine; venlafaxine alone

SUMMARY:
The purpose of this study is to evaluate the efficacy of repetitive transcranial magnetic stimulation in the prevention of relapse of the symptoms of depression. Primary Outcome Measures:Time between subject randomization to treatment and the first occurrence of a relapse during the Relapse Prevention Period. Secondary Outcome Measures: Symptom change as measured by Hamilton Depression Rating Scale (HDRS); Illness severity change as measured by Clinical Global Impression of Severity for depression(CGI-S-DEP); Change in subject functioning using the Personal and Social Performance Scale.

DETAILED DESCRIPTION:
Transcranial magnetic stimulation is a noninvasive technique that can influence specific areas of the brain and has very few side effects.Several factors characterize repetitive transcranial magnetic stimulation (rTMS) as a strategic aid in the treatment of depression.Depression is a chronic illness and generally requires life-long treatment. However, up to current days there have been no studies evaluating the effects of rTMS in the maintenance treatment of depression. This is a randomized, double-blind, placebo-controlled, parallel-group, multicenter study to evaluate the efficacy of rTMS, as monotherapy, relative to placebo in delaying the time to relapse in patients with depression. Patients with acute symptoms of depression will be enrolled. The study will consist of 4 periods: an up to 7 days screening/tolerability period, a 6-week open-label flexible dose lead-in period, a 6-week open-label fixed dose stabilization period, and a 12 months double-blind relapse prevention period. The study will consist of 4 phases: a screening/tolerability phase of up to 7 days; an open-label, flexible-dose lead-in phase of 8 weeks; an open-label, fixed-dose stabilization phase of 6 weeks; and a single-blind relapse prevention phase of 12 months. During the open-label phase, all patients will be treated with venlafaxine. Remitterswith Hamilton Rating Scale for Depression [HAM-D17] score ≤ 7will be eligible to enter the single-blind phase and will be randomly assigned to one of three groups: group 1 on active rTMS and venlafaxine; group 2 on sham rTMS and venlafaxine; group 3 on venlafaxine alone. Efficacy will be evaluated during the study using relapse assessment (time between subject randomization to treatment and the first occurrence of relapse). Secondary outcome measures will include: symptom changes, measured by the Hamilton Rating Scale for Depression [HAM-D17]; illness severity changes, measured by the Clinical Global Impression of Severity for Depression (CGI-S-DEP); and changes in subject functioning, assessed with the Personal and Social Performance Scale. Safety will be assessed throughout the study by monitoring of adverse events, clinical laboratory tests, electrocardiography, and measurements of vital signs (temperature, pulse and blood pressure) and weight. Suicidality will be assessed by the Columbia Suicide Severity Rating Scale (C-SSRS). A 10 milliliter pharmacogenomic blood sample (sample for DNA research) will be collected from patients who give separate written informed consent for this part of the study.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of depression
* Experiencing an acute exacerbation of depression symptoms
* Baseline score of at least 14 points on the Hamilton Depression rating Scale-17 items
* Healthy based on physical examinations, electrocardiogram (ECG), laboratory tests, medical history, and vital signs measurements

Exclusion Criteria:

* Comprised ferromagnetic metallic implants
* Pacemakers
* Previous neurosurgery
* History of seizures
* Major head trauma
* Alcoholism
* Drug addiction
* Any psychiatric or neurological disorder other than depression and anxiety
* Psychotic depression
* Suicidal propensities

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 391 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2017-02-25 (Actual)

PRIMARY OUTCOMES:
Time for relapse | Participants will be followed for the duration of 15 month double-blind Relapse Prevention Period, an expected average of 5 weeks
  Time between subject randomization to treatment and the first occurrence of a relapse during the Relapse Prevention Period

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale | baseline and 15 months
  Reduction on the scores of HDRS (as on the scores of Depression Scale and Hamilton Anxiety Scale; and improves the global clinical status in Clinical Global Impression, Global Assessment Scale and 36-item Short-form Health Survey - Quality of Life)
Illness severity change | baseline and 15 months
  Illness severity change as measured by Clinical Global Impression of Severity for depression.
subject functioning | baseline and 15 months
  Change in subject functioning using the Personal and Social Performance Scale (PSP)

CONTACTS AND LOCATIONS:
Locations (1):
- Qingrong, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Wang H, Xue Y, Chen Y, Zhang R, Wang H, Zhang Y, Gan J, Zhang L, Tan Q. Efficacy of repetitive transcranial magnetic stimulation in the prevention of relapse of depression: study protocol for a randomized controlled trial. Trials. 2013 Oct 17;14:338. doi: 10.1186/1745-6215-14-338. PMID 24135054